CLINICAL TRIAL: NCT06669897
Title: Validation of a Questionnaire to Measure Cough Severity in Patients With Chronic Cough
Brief Title: Validation of a Questionnaire to Measure Cough Severity
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TOS-2023-133
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-10

CONDITIONS: Cough
Keywords: Cough; Chronic cough
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Chronic cough
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Chronic cough questionnaire

SUMMARY:
To design and validate a questionnaire that allows objective assessment of the severity of chronic cough

DETAILED DESCRIPTION:
Chronic cough is a common disease that has important consequences for patients, ranging from physical to psychological and social aspects. However, there is currently no tool to objectively validate cough severity.

The aim of the study is to design and validate a questionnaire to objectively assess the severity of chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 99 years
* Clinical diagnosis of chronic cough or healthy volunteers
* Good understanding of Spanish

Exclusion Criteria:

* Non-Spanish-speaking patients
* Inability to complete the questionnaires
* Failure to sign the informed consent form

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spanish-speaking patients with previous diagnosis of chronic cough or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
A questionnaire for assessing the severity of chronic cough | 1 year
  To design and validate a questionnaire to objectively assess the severity of chronic cough

SECONDARY OUTCOMES:
Correlation of the results of the questionnaire with frequency of cough | 1 year
  Perform a statistical analysis to determine the correlation of the results of the questionnaire with frequency of cough

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo-Lessmann, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (6):
- Spain (6):
  - Hospital Universitario Hermanos Trias y Pujol, Badalona, Barcelona
  - Hospital Univesitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] French CT, Irwin RS, Fletcher KE, Adams TM. Evaluation of a cough-specific quality-of-life questionnaire. Chest. 2002 Apr;121(4):1123-31. doi: 10.1378/chest.121.4.1123. PMID 11948042
- [Background] McGarvey L, Gibson PG. What Is Chronic Cough? Terminology. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):1711-1714. doi: 10.1016/j.jaip.2019.04.012. Epub 2019 Apr 17. PMID 31002958
- [Background] Morice AH, McGarvey LP, Dicpinigaitis PV. Cough hypersensitivity syndrome is an important clinical concept: a pro/con debate. Lung. 2012 Feb;190(1):3-9. doi: 10.1007/s00408-011-9351-y. Epub 2011 Dec 22. PMID 22186805
- [Background] Haque RA, Usmani OS, Barnes PJ. Chronic idiopathic cough: a discrete clinical entity? Chest. 2005 May;127(5):1710-3. doi: 10.1378/chest.127.5.1710. PMID 15888850
- [Background] Song WJ, Chang YS, Faruqi S, Kim JY, Kang MG, Kim S, Jo EJ, Kim MH, Plevkova J, Park HW, Cho SH, Morice AH. The global epidemiology of chronic cough in adults: a systematic review and meta-analysis. Eur Respir J. 2015 May;45(5):1479-81. doi: 10.1183/09031936.00218714. Epub 2015 Feb 5. No abstract available. PMID 25657027
- [Background] Morice A. Chronic cough: epidemiology. Chron Respir Dis. 2008;5(1):43-7. doi: 10.1177/1479972307084252. PMID 18303101
- [Background] Irwin RS, Baumann MH, Bolser DC, Boulet LP, Braman SS, Brightling CE, Brown KK, Canning BJ, Chang AB, Dicpinigaitis PV, Eccles R, Glomb WB, Goldstein LB, Graham LM, Hargreave FE, Kvale PA, Lewis SZ, McCool FD, McCrory DC, Prakash UBS, Pratter MR, Rosen MJ, Schulman E, Shannon JJ, Hammond CS, Tarlo SM. Diagnosis and management of cough executive summary: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):1S-23S. doi: 10.1378/chest.129.1_suppl.1S. No abstract available. PMID 16428686